CLINICAL TRIAL: NCT06532500
Title: I-CARE: A Pilot Study of Cognitive Behavioural Therapy(CBT) for Mood and Anxiety Disorders
Acronym: I-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Mark Sinyor, Staff Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6352
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mood Disorders; Anxiety Disorders
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants have a 50/50 chance of being assigned to the CBT-MyOWL or CBT-as-usual group for 12 sessions of either therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-MyOWL (Experimental): A novel talk therapy model where we incorporate the standard CBT model with experiential learning while reading the third novel in the Harry Potter series to teach coping skills and emotional resiliency. The 12 sessions of CBT-MyOWL will follow a modestly adapted version of the intervention offered on www.myowl.org. The therapist will cover topics such as risk and protective factors for distress and mental health problems, cognitive distortions, cognitive reframing, fear hierarchies, behavioural activation and core beliefs while reading Harry Potter and the Prisoner of Azkaban.
  Interventions: Behavioral: CBT-MyOWL
- CBT-as-usual (Active Comparator): A talk therapy where participants will be encouraged to recognize distortions in thinking and then to reevaluate them in light of the evidence, gain a better understanding of how their behaviour contributes to wellbeing, learn to use problem-solving skills to cope with difficult situations, and learn to develop a greater sense of confidence in one's own abilities. This is the control group, and they will be utilizing the 'Mind over Mood' and/or the 'Anxiety and Phobia Workbook' according to the primary diagnosis.
  Interventions: Behavioral: CBT-as-usual

INTERVENTIONS:
Behavioral: CBT-MyOWL — 12-sessions of CBT-MyOWL
  Arms: CBT-MyOWL
Behavioral: CBT-as-usual — 12-sessions of CBT using Mind Over Mood or Anxiety Phobia
  Arms: CBT-as-usual

SUMMARY:
The goal of this clinical trial is to learn if CBT(Cognitive Behavioural Therapy)-MyOWL(Optimizing Wellness through Literature) is feasible, leads to better patient retention, and has high acceptability by youth psychiatric outpatients with mood and/or anxiety disorder aged 14-19. The main questions it aims to answer are:

Primary Objective (feasibility): To determine whether a clinically meaningful proportion of youth complete a full course of CBT-MyOWL / CBT-as-usual.

Primary Objective (acceptability): To determine whether the CBT-MyOWL and CBT-as-usual interventions delivered are acceptable to youth participants.

Secondary Objectives:

1. To determine whether CBT-MyOWL enhances time of retention compared to CBT-as-usual.
2. To determine whether youth who receive CBT-MyOWL have improved scores on all of the following over the course of treatment and endpoint compared to youth who receive CBT-as usual: i) depression and anxiety ii) suicidal ideation, iii) self-harm, and iv) coping and emotional resiliency.

Participants will:

Participate in 12 sessions of either CBT-MyOWL or CBT-as-usual (active control) Completes 4-5 questionnaires at sessions 3,6,9,12 Complete the acceptability and exit interview at session 12

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-19
* Primary diagnosis of a mood disorder or an anxiety disorder
* Ability to understand written and spoken English and to read a novel
* Treating physician considers CBT as indicated for the patient

Exclusion Criteria:

* Patients already participating in active CBT therapy or recently completed CBT treatment (within the past 3 months)
* Active psychosis or mania

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Dropout rates | Comparing the baseline and across the 12 weeks
  To determine whether a clinically meaningful proportion of youth complete a full course of CBT-MyOWL / CBT-as-usual.
Acceptability Questionnaire | 12 week session
  To determine whether the CBT-MyOWL and CBT-as-usual interventions delivered are acceptable to youth participants.*
  *Note, given that CBT-as-usual is the gold standard treatment, we assume it will be feasible and acceptable and are mainly interested in the feasibility and acceptability of CBT-MyOWL. However, we believe it is important to measure both and will report on any differences identified.

SECONDARY OUTCOMES:
Retention | Comparing the baseline and across the 12 weeks
  To determine whether CBT-MyOWL enhances time of retention compared to CBT-as-usual.
Change from Baseline in Revised Children's Anxiety and Depression Scale score to weeks 3, 6, 9 and 12 | Baseline, Week 3, Week 6, Week 9 and Week 12
  The Revised Children's Anxiety and Depression Scale (RCADS) is a 25-item self-report designed to measure anxiety and depression.
  The total score of the RCADS-25 is calculated by assigning 0-3 to the response categories of "never", "sometimes", "often", "always", respectively. The sum of all 25 items is tallied and represents the severity of general anxiety and depressive symptoms. The minimum score is 0 and the maximum score is 75. Higher scores mean a worse outcome.
  Converted scores on the total scale and both sub-scales are divided into scoring ranges, where: (a) scores below 65 represent low severity, (b) scores between 65-70 represent medium severity and are on the borderline clinical threshold, and (c) scores above 70 represent high severity and are above the clinical threshold.
Change from Baseline in The Coping Scale for Children and Youth score to weeks 3, 6, 9 and 12 | Baseline, Week 3, Week 6, Week 9 and Week 12
  The Coping Scale for Children and Youth (CSCY) is a 29-item self-report designed to measure coping behaviours.
  The total score of the CSCY is calculated by assigning 0-3 to the response categories of "never", "sometimes", "often", and "very often", respectively. The minimum score is 0 and the maximum score is 29. Higher scores mean a better outcome.
Change from Baseline in The Cognitive and Behavioural Response to Stress Scale score to weeks 3, 6, 9 and 12 | Baseline, Week 3, Week 6, Week 9 and Week 12
  The Cognitive and Behavioural Response to Stress Scale (CB-RSS) is a 19-item self-report designed to measure cognitive and behavioural responses in a stressful situation. 0 = Never, 1 = Rarely, 2 = Occasionally, 3 = Sometimes, 4 = Often, 5 = Very often, 6 = Always. Higher scores means a better outcome.
Changes from Baseline in The Columbia-Suicide Severity Rating Scale score to weeks 3, 6, 9 and 12 | Baseline, Week 3, Week 6, Week 9 and Week 12
  The Columbia-Suicide Severity Rating Scale (CSSRS) is a 6-item research assistant/coordinator-rated questionnaire. Our research team also added one item on non-suicidal self-injurious behaviour. The outcome is measured by comparing the number of times the participants in the CBT-MyOWL versus the CBT-as-usual group answered yes/no to the self-harm behaviour question throughout the four times asked during the CBT.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sinyor, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No